CLINICAL TRIAL: NCT05626387
Title: Mycophenolate Mofetil and Prednisolone Versus Prednisolone Alone in Fibrotic Hypersensitivity Pneumonitis: a Randomized Controlled Trial
Brief Title: An RCT of Mycophenolate Mofetil (MMF) in Fibrotic Hypersensitivity Pneumonitis
Acronym: MYCOHYPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYCOHYPE
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Hypersensitivity Pneumonitis
Keywords: HP; interstitial lung disease; ILD; diffuse parenchymal lung disease
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic; Lung Diseases, Interstitial | interventions — Mycophenolic Acid; Prednisolone; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone alone (Active Comparator): Oral prednisolone will be administered over 52 weeks, according to following schedule 0.75 mg/kg x 2 weeks 0.5 mg/kg x 2 weeks 20 mg/day x 4 weeks 15 mg/day x 4 weeks 10 mg/day x 4 weeks 5 mg/day x 10 weeks 5 mg on alternate days x 26 weeks
  Interventions: Drug: Prednisolone
- Mycophenolate mofetil plus prednisolone (Experimental): Oral prednisolone will be administered according to the schedule in the prednisolone alone arm. Mycophenolate mofetil will be administered starting from 2 weeks after randomization. It will be initiated at a dose of 500 mg twice daily and will be escalated to 1000 mg twice daily after two weeks.
  Interventions: Drug: Mycophenolate Mofetil plus prednisolone

INTERVENTIONS:
Drug: Mycophenolate Mofetil plus prednisolone — Prednisolone is a glucocorticoid that suppresses inflammation by several mechanisms. Mycophenolate mofetil (MMF) is an immunosuppressive drug that acts by inhibiting the proliferation of T-lymphocytes and suppressing the recruitment of lymphocytes and monocytes into the sites of inflammation.
  Other Names: Intervention
  Arms: Mycophenolate mofetil plus prednisolone
Drug: Prednisolone — Prednisolone is a glucocorticoid that suppresses inflammation by several mechanisms.
  Other Names: Control
  Arms: Prednisolone alone

SUMMARY:
To our knowledge, there is no randomized controlled trial assessing the efficacy of mycophenolate mofetil (MMF) in the treatment of HP. We aim to perform a randomized study to assess the efficacy and safety of a regimen consisting of MMF and prednisolone against a regimen consisting of prednisolone alone for treating fibrotic HP. We hypothesize that the treatment of patients with fibrotic HP with MMF and prednisolone will be more effective and safer than treatment with prednisolone alone.

DETAILED DESCRIPTION:
Hypersensitivity pneumonitis (HP) is a complex immunologically-mediated interstitial lung disease (ILD) resulting from sensitization to an inhaled antigen. It may be categorized into acute (acute/subacute) or chronic forms based on the duration of disease or evidence of chronicity on radiological or pathological findings. Lately, the American Thoracic Society (ATS) Guidelines 2020 has endorsed a new classification of HP into non-fibrotic and fibrotic types based on the absence or presence of signs of fibrosis on chest computed tomography (CT) or histology. According to a survey study, about three-fourths of respiratory physicians believe that fibrotic HP should be treated with glucocorticoids as the treatment of first choice, which also reflects the practice in most centers worldwide. However, there is some evidence that glucocorticoids may not be effective in the long-term treatment of fibrotic HP. Also, glucocorticoids are associated with several adverse effects especially when used over a long duration. Therefore, most experts recommend that glucocorticoids should be tapered to the lowest possible dose after a trial of about three months in chronic/fibrotic HP.

Hypersensitivity pneumonitis is characterized by an exaggerated T cell-mediated immune inflammatory response (T-lymphocytic alveolitis) due to increased migration, local proliferation, and decreased programmed cell death of lymphocytes. Mycophenolate mofetil (MMF) is an immunosuppressive drug that acts by inhibiting the proliferation of T-lymphocytes and suppressing the recruitment of lymphocytes and monocytes into the sites of inflammation. Therefore, MMF is likely to be effective in the treatment of HP. There are only a few retrospective studies on the efficacy of MMF in the treatment of HP. To our knowledge, there is no randomized controlled trial assessing the efficacy of MMF in the treatment of HP.

We aim to perform a randomized study to assess the efficacy and safety of a regimen consisting of MMF and prednisolone against a regimen consisting of prednisolone alone for treating fibrotic HP. We hypothesize that the treatment of patients with fibrotic HP with MMF and prednisolone will be more effective and safer than treatment with prednisolone alone.

ELIGIBILITY:
Inclusion Criteria:

i. A diagnosis of fibrotic hypersensitivity pneumonitis according to the criteria proposed in the American Thoracic Society Guideline 2020 ii. Screening FVC at least 40% of the predicted value iii. Able to provide a written, informed consent for participation in the trial

Exclusion Criteria:

i. Baseline FVC <40% predicted ii. Leucopenia (white blood cell count <4·0 × 10^9 per L), significant thrombocytopenia (platelet count <100 × 10^9 per L), or clinically significant anemia (hemoglobin <10 g/dL) iii. Baseline liver transaminases (alanine aminotransferase and aspartate aminotransferase) or bilirubin more than 1·5 times the upper normal limit (except in the case of Gilbert's syndrome) iv. Serum creatinine higher than 2.0 mg/dL v. Uncontrolled congestive heart failure vi. Receipt of prednisolone (more than or equal to 10 mg/day, or equivalent), in the 4 weeks before randomization vii. Prior use of prednisolone (more than or equal to 10 mg/day, or equivalent), MMF, azathioprine, cyclophosphamide, cyclosporine or any other non-glucocorticoid immunosuppressant drug, or antifibrotic agents for more than 12 weeks in the previous year viii. Active infection (lung or elsewhere) whose management would be compromised by MMF or prednisolone ix. Other serious concomitant medical illness (eg, cancer), chronic debilitating illness (other than chronic HP), or drug abuse x. Pregnancy (documented by urine pregnancy test) or breastfeeding xi. Unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-10-23 (Estimated)

PRIMARY OUTCOMES:
Lung function (FVC) decline | 52 weeks
  Annual rate of decline in forced vital capacity (FVC) assessed using spirometry assessed over 52 weeks

SECONDARY OUTCOMES:
FEV1 decline | 52 weeks
  Annual rate of decline in forced expiratory volume in one second (FEV1) assessed using spirometry over 52 weeks
Severity of breathlessness | 52 weeks
  Severity of dyspnea as assessed using the modified Medical Research Council (mMRC) scale
Six-minute walk distance | 52 weeks
  Change in six-minute walk distance (6MWD) from the baseline that will be performed using American Thoracic Society guidelines
Disease specific health status | 52 weeks
  Interstitial lung disease (ILD)-specific health status as assessed by the King's Brief ILD Questionnaire
Diffusion capacity | 52 weeks
  Change in the diffusion capacity for carbon monoxide (DLCO) of the lung from the baseline
Proportion of subjects who develop progressive pulmonary fibrosis (PPF) | 52 weeks
  Proportion of subjects who develop progressive pulmonary fibrosis (PPF), which will be defined using the American Thoracic Society 2022 recommendations
Proportion of subjects who develop acute exacerbation(s) | 52 weeks
  Proportion of subjects who develop acute exacerbation(s), which will be defined using the definition proposed by the International Working Group in 2016
Treatment-emergent adverse effects | 52 weeks
  Number of treatment-related adverse effects in each arm. The grading of adverse events according to the Common Terminology Criteria for Adverse Events version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Sahajal Dhooria, MD, DM, Principal Investigator — Postgraduate Institute of Medical Education and Research, Chandigarh, India
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data might be made available on request, after the completion of the study
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the completion and publication of the study results
Access Criteria: On a reasonable request